CLINICAL TRIAL: NCT02161497
Title: Comparison of Clinical History Taking Versus the Addition of an Electronic Patient File Consultation in Pediatric Pre-operative Assessments
Brief Title: Clinical History Taking Versus the Addition of an Electronic File Consultation in Pediatric Pre-operative Assessments
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0313-13-MMC
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-06

CONDITIONS: Anesthesia
Keywords: Medical History Taking; Electronic Health Records; Pediatrics; Parents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are studying the difference between the history taken from parents prior to their child's anesthesia to information gleaned routinely from a patient information system called Ofek.

DETAILED DESCRIPTION:
Introduction One of the cornerstones of pre-operative assessment is an accurate clinical history. In pediatric anesthetic practice, the history is typically obtained from an accompanying parent. A letter from the patient's primary care physician may accompany the child for elective cases, but typically contains general information and may omit recent illnesses. In addition, parents may underplay or deny respiratory problems such as upper or lower respiratory tract infections, asthma, cough or snoring as the norm for a particular child and not understand their importance in pre-operative assessment.

The Clalit Health Services HMO is Israel's largest health insurer and has a comprehensive online patient database for healthcare workers to use for patient care. The Ofek patient electronic record system allows the physician to view patient community and hospital records, including special investigations and drug prescription and purchases, updated in real time. Recently, the system was upgraded to view patient records from all of the four Israeli HMOs. This has enabled the treating physicians' electronic record access to any patient that may present.

The investigators see this development as a major advantage. Moreover, in the pediatric pre-anesthetic assessment setting, the clinical history may be verified by the Ofek system.

Aim To compare the details obtained at pre-anesthetic clinical history given by parents of children undergoing surgery to those obtained using the Ofek electronic patient record system. In addition, we would like to inquire into the reasons that discrepancies may exist between clinical histories and the electronic patient record and the clinical impact of those differences on clinical decision making.

Methods Two hundred children and parent/s will undergo pre-anesthetic clinical history taking. Each parent and child will be screened pre-operatively by a senior anesthesiology resident using the Meir Medical Center Anesthesia pre-operative pediatric assessment form. Thereafter, the resident will open the electronic patient file using the Ofek system and additional information, if present will be noted. Parents will be asked, where relevant, for the reason additional information gleaned via Ofek was omitted during the direct questioning. If the clinical history and/or Ofek resulted in changes in patient management, this will be noted as well.

Data to be collected will include the number of discrepancies between clinical history and information obtained using Ofek and the reasons for those differences will be noted. In addition, the source of all information whether obtained via clinical history or Ofek will be noted. If information obtained by either of the abovementioned means results in changes in clinical management, these will be noted as well. The data collected from parents and Ofek is done so without any connection to the study.

Statistical analysis Comparisons between nominal variables will be analyzed by Chi-Square and derivatives of it (McNemar, Kappa). Continuous parameters - by paired tests -parametric and non-parametric,each as appropriate. Reliability between "Ofek" and clinical history will be measured by Intra-Class Coefficients and coefficient of variations (CoV). All statistical procedures, each as needed.

ELIGIBILITY:
Inclusion Criteria:

* Children presenting with parent/s for pre-operative assessment
* Ages newborn to 16 years
* Elective and emergency surgery

Exclusion Criteria:

* Premature infants still hospitalized in the Neonatal intensive care unit

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parents of children being interviewed at pre anesthesia assessment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of discrepancies found between clinical history and information received from OFEK system, the reasons for those discrepancies and how they influenced peri-operative clinical decision making. | Immediate

SECONDARY OUTCOMES:
Average time spent using OFEK system per patient. | Immediate
Average time spent taking clinical history per patient. | Immediate
Number of discrepancies found between clinical history and information received from OFEK system that do not influence peri-operative clinical decision making. | Immediate
Reasons for each discrepancy. | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: David R Hoppenstein, MBBCh, Principal Investigator — Meir Medical Center Tel Aviv University
Locations (1):
- Meir Medical Center, Kfar Saba, Israel